CLINICAL TRIAL: NCT04277195
Title: Developing a Diagnostic Tool, Using SPAG5, for Predicting Clinical Benefit From Standard Anthracycline Combination (AC) in Breast Cancer
Brief Title: Developing a Diagnostic Tool to Predict Response to Chemotherapy
Acronym: SPAG5
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Nottingham University Hospitals NHS Trust (Other)
Collaborators: University of Nottingham (Other); Nottingham Trent University (Other); University of Lincoln (Other)
Responsible Party: Sponsor
Other Study IDs: 18ON009; II-LA-0417-20004 (Other Grant/Funding Number: National Institute for Health Research); 2125 (Other Grant/Funding Number: Nottingham Hospitals Charity)
Record Dates: First submitted 2019-11-18; First posted 2020-02-20 (Actual); Last update posted 2020-02-20 (Actual); Status verified 2019-11

CONDITIONS: Breast Cancer
Keywords: Breast Cancer; SPAG5; Chemotherapy; Anthracycline; Predictive test; Predictive assay; SPerm associated AntiGen 5; ASTRIN
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — All tissue used in this study will be stored material which was collected from patients as part of their standard treatment for breast cancer. No new tests or samples are required. This tissue is preserved in a wax block in the hospital pathology archives. It is standard practice at the hospital for patients to consent for any excess tissue, not required for diagnostic purposes, to be left available for use in research. These blocks will be collected and assessed. Those which still have sufficient tissue can be cut in to thin sections (4µm) and stained in the lab to test for the presents of proteins which are important in cancer biology.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- NUH Adjuvant Breast Cancer Cohort: Historical: This is a series of breast cancer patients treated with adjuvant therapy, who were identified and samples selected for inclusion in the Nottingham Tenovus Breast research project by Prof Ian Ellis's research group (1986-1999; n=1650). The clinical dataset for this cohort of breast cancer patients has been collected in a master clinical database by the team supporting Professor Ian Ellis. The study research team will work with a pseudo-anonymised copy of this dataset.
  Interventions: Diagnostic Test: SPAG5 Assay
- NUH Adjuvant Breast Cancer Cohort: New: A series of breast cancer patients treated with adjuvant therapy, who were identified and samples selected for inclusion in the Nottingham Tenovus Breast research project by Prof Ian Ellis's research group (2000-2006; n=2000). The clinical dataset for this cohort of breast cancer patients has been collected in a master clinical database by the team supporting Professor Ian Ellis. The study research team will work with a pseudo-anonymised copy of this dataset.
  Interventions: Diagnostic Test: SPAG5 Assay
- NUH Neoadjuvant Breast Cancer Cohort: For many years clinical data on this cohort of breast cancer patients has been collected in a master clinical database by the clinical team supporting Dr Chan (1996-2021; n=900 patients). This has been used for internal audits and reviews of clinical practice. The study research team will work with a pseudo-anonymised copy of this dataset.
  Interventions: Diagnostic Test: SPAG5 Assay
- NUH Oncotype DX tested Adjuvant Breast Cancer Cohort: A list of patients tested with Oncotype DX as part of their standard treatment pathway (2015-2021; n=200) will be collected and will form the basis of a master clinical database for this cohort. The database will be managed and populated by the clinical team supporting Dr Chan. The study research team will work with a pseudo-anonymised copy of this dataset.
  Interventions: Diagnostic Test: SPAG5 Assay

INTERVENTIONS:
Diagnostic Test: SPAG5 Assay — Testing for SPAG5 expression in the tumour.

SUMMARY:
Every year nearly 62,000 people are diagnosed with breast cancer in the UK. One in eight women in the UK will develop breast cancer in their lifetime.

The investigators are developing an inexpensive test to accurately predict how breast cancer patients will respond to the standard chemotherapy Anthracycline (AC). Only 15-20% of patients have no tumour remaining following AC, so a method of treatment selection is urgently needed.

Breast cancers are currently treated with a combination of chemotherapy, targeted therapy and surgery. However, breast cancers are not identical; each tumour's individual characteristics affect how they respond to treatment. Recently the investigators discovered a new tumour characteristic, a protein which is unusually active in approximately 20% of breast cancers. It was found that a patient whose tumour showed high activity often respond well to AC, and vice versa.

AC is an aggressive treatment which can potentially cause severe side effects, including a risk of permanent heart damage. It is important, therefore, to spare those patients who will not benefit from AC the physical and emotional side-effects of this drug. Currently, there is no predictive test for selecting which patients will benefit from AC and which will not. The investigators have shown that an accurate prediction can be made by testing the activity of a protein called 'SPerm associated AntiGen 5' (SPAG5) in tumour tissue.

The aim is to develop a clinical SPAG5 testing kit that can be used by hospital laboratories to determine the activity of SPAG5 in the tumour. This information will help guide the choice of treatment and achieve better patient outcomes.

In June 2018 the investigators started a three year National Institute for Health Research (NIHR) funded project to develop a lab test that could form the basis of a SPAG5 testing kit.

DETAILED DESCRIPTION:
Approximately 16,700,000 people are diagnosed with breast cancer (BC) worldwide each year, with 500,000 people dying annually. In the UK alone, each year nearly 62,000 people are diagnosed with BC, with one in eight women developing BC in their lifetime. Breast cancers are currently treated with a combination of chemotherapy, targeted therapy and surgery. However, breast cancers are not identical; each tumour's individual characteristics affect how they respond to treatment. In many cases, treatment options are limited and patients are often given sub-optimal treatments which are associated with burdensome side effects. For instance, despite chemotherapy being offered to about 60-70% of patients with BC, either alone or in combination with other targeted therapies, results from a meta-analysis of 123 randomised trials including more than 100,000 patients has shown that chemotherapy reduces recurrence and mortality in only 20 to 33% of patients. Therefore, 80-67% of patients endured this aggressive chemotherapy treatment and did not benefit; unnecessarily suffering the serious physical and emotional side effects, including a risk of permanent heart damage. Currently, there is no predictive test for selecting which patients will benefit from receiving chemotherapy and which will not.

In clinical practice, the decision to use chemotherapy or not depends on evaluating the risk of recurrence and prognosis by interpreting prognostic clinicopathological features including high cost multi-gene tests such as Oncotype DX (Genomic Health Inc.), Mamma-Print (Agendia), and PAM50 (NanoString). Unfortunately, almost all these molecular approaches share common issues, such as insufficiently high levels of evidence, overfitting of computational models, and high false discovery rates. Furthermore, they might not be available for clinical, logistical or financial reasons. Therefore, there is an urgent need for a cost effective, reliable, sensitive, specific, validated biomarker based approach for optimising chemotherapy treatments in patients with BC.

Recently, the investigators have shown that an accurate prediction can be made by testing the activity of a protein called 'SPerm associated AntiGen 5' (SPAG5) in tumour tissue. In a study, published in Lancet Oncology (2016), the investigators showed that SPAG5 gene amplification, as well as SPAG5 transcript and SPAG5 protein overexpression, were all associated with poor clinical outcome, and were independent predictors for chemotherapy response.

The prognostic and predictive power of SPAG5 outperforms many currently used tests including: the standard cancer proliferation index (Ki67), prognostic clinicopathological factors such as the American Joint Committee on Cancer (AJCC) stage and Nottingham Prognostic Index, as well as other currently available multigene-tests including PAM-50, 96-gene genomic grade index, Genomic Chemo Sensitivity Predictor, the Diagonal Linear Discrimination Analysis of 30-gene signature, and the Adjuvant Online index.

The most immediately useful aspect of our original findings is the potential ability to distinguish those patients with BC who are likely to benefit from standard Anthracycline combination (AC) chemotherapy regimens from those who will not. Therefore our findings have the potential to deliver an accurate predictive biomarker for chemotherapy response in BC which would enable the effective tailoring of treatment to the individual patient. Furthermore, the analysis of SPAG5 expression could underpin the development of novel strategies for more effective management and treatment of the disease.

The work undertaken by the investigators on SPAG5 testing has relied on a commercially available polyclonal antibody (PAb) against SPAG5 marketed by Sigma Aldrich and produced by Atlas Antibodies. This has a number of problems when aiming to develop a SPAG5 based clinical test. Firstly, a PAb is a mixture of antibodies and so it lacks specificity and sensitivity. Also, as a PAb it is extracted directly from an animal, constraining the supply and placing a finite limit on the availability of the antibody, as the animal will die one day ending our ability to provide the test. Thirdly, the PAb is owned by a company and so the cost and availability of any test will be subject to that company's decision. Therefore it is essential to develop a monoclonal antibody (MAb) that is suitable for immunohistochemistry staining of Formalin Fixed Paraffin Embedded (FFPE) tissue.

To overcome these problems the investigators chose to develop a SPAG5 targeting MAb that can be taken through the evaluation, clinical testing and regulatory approval process to become a SPAG5 clinical test. Moreover, once the MAb is developed, the validation of previous results will be carried out on a large number of BC cases to verify the prognostic and predictive powers of the antibody. In addition, the predictive utility for chemo-sensitivity of SPAG5 MAb and PAb will be compared to each other and to rival Immunohistochemistry (IHC) tests such as Ki67 and the rival gene expression tests. A bespoke gene panel will be developed for the nanoString nCounter™ FLEX instrument, featuring genes used in PAM-50, 21-gene recurrence Genomic-Chemo-Sensitivity-Predictor, and the 30-gene-DLDA tests, alongside SPAG5 and Ki67.

In June 2018 the investigators were granted funding to pursue this work by the NIHR Invention for innovation grant program.

ELIGIBILITY:
Inclusion Criteria:

* Histological diagnosis of primary invasive breast cancer.
* Any hormone receptor status (Oestrogen Receptor, Progesterone Receptor).
* Any Human epidermal growth factor receptor 2 (HER2) receptor status.
* 18 to 90 years old.

Exclusion Criteria:

* Histological diagnosis of any other cancer type.
* Evidence of distant metastatic disease at diagnosis.
* Insufficient tumour tissue available for research use in tissue blocks held in the NUH Trust pathology archive.
* Outside of stated inclusion age range.

Ages: 18 Years to 90 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This is a retrospective study, involving patients diagnosed with breast cancer. For each patient cohort featured in the study plan we will be using archived patient samples collected as part of each patients standard care pathway. At no point are patients prospectively recruited to the study. Many of these cohorts have already been assembled as part of past projects to construct Tissue Micro Array's (TMA).
Sampling Method: Probability Sample
Enrollment: 4750 (Estimated)
Dates: Start 2019-11-07 (Actual); Primary Completion 2021-05-31 (Estimated); Study Completion 2021-05-31 (Estimated)

PRIMARY OUTCOMES:
Production of a SPAG5 assay | 3 years
  The primary objective of the study is to deliver a new monoclonal antibody based test that can be used to measure the level of the SPAG5 protein in FFPE breast cancer samples. This objective will only be reached if the new antibodies statistical power, to predict response of breast cancer to chemotherapy, equals or exceeds that of the commercial research grade antibody used in our past publications.
  The response end points for adjuvant treatment (Surgery then Chemotherapy) will be Relapse Free Survival and Breast Cancer Specific Survival, at 5 and 10 years post treatment. The response end point for neoadjuvant treatment it will be pathological Complete Response at surgery.
  The delivery of this test will lead to the development of a clinical testing kit that can be used by hospital laboratories, to help guide the choice of treatment and achieve better patient outcomes.

SECONDARY OUTCOMES:
Testing of the SPAG5 assay against rival genetic tests | 3 years
  To test this new antibody against the rival genetic tests that have been published in the literature, as well as the few which have begun to be used in the clinic, to determine the advantages and disadvantages of each in predicting response to treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- Nottingham University Hospitals NHS Trust, Nottingham, Nottinghamshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Abdel-Fatah TMA, Agarwal D, Liu DX, Russell R, Rueda OM, Liu K, Xu B, Moseley PM, Green AR, Pockley AG, Rees RC, Caldas C, Ellis IO, Ball GR, Chan SYT. SPAG5 as a prognostic biomarker and chemotherapy sensitivity predictor in breast cancer: a retrospective, integrated genomic, transcriptomic, and protein analysis. Lancet Oncol. 2016 Jul;17(7):1004-1018. doi: 10.1016/S1470-2045(16)00174-1. Epub 2016 Jun 14. PMID 27312051
- See also: NIHR funding and awards, research award details — https://fundingawards.nihr.ac.uk/award/II-LA-0417-20004